CLINICAL TRIAL: NCT03531203
Title: The Effect of Soursop Supplementation on Blood Pressure, Serum Uric Acid and Kidney Function in Prehypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Mlati Study Group, Faculty of Medicine, Gadjah Mada University (Unknown)
Responsible Party: Principal Investigator, Mochammad Sja'bani, Professor, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soursop Supplementation 2017
Record Dates: First submitted 2018-04-26; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Blood Pressure; Prehypertension; Uric Acid
Keywords: soursop; supplementation; prehypertension; uric acid; randomized controlled trial
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Soursop (Experimental): Treatment group (with soursop group) was a group which receive soursop supplementation
  Interventions: Dietary Supplement: Soursop supplementation
- Without Soursop (Placebo Comparator): Control group (without soursop group) was a group which do not receive any intervention (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Soursop supplementation — The soursop supplementation was given to treatment group (with soursop group) 2 times a day for 100 g each for 3 months period.
  Arms: With Soursop
Other: Placebo — Control group (without soursop group) was left without treatment during study period
  Arms: Without Soursop

SUMMARY:
This study was a randomized controlled trial study. The aim of this study was to determine the effect of soursop fruit supplementation on blood pressure (BP), serum uric acid (SUA), and kidney function.

The definition of prehypertension and hypertension was accepted as delivered in The Seventh Report of the Joint National Committee (JNC 7) as the systolic BP was 120 - 139 mmHg and diastolic BP was 80 - 89 mmHg for prehypertension, while systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg for hypertension.

Based on the study by Sja'bani (2014), the cut-off point of (SUA) was divided into 3 categories, which are normal (< 5 mg/dL), high-normal (5 - <7 mg/dL), and high (≥ 7 mg/dL).

A number of 143 people with essential prehypertension and high normal uric acid level were assigned as subject in this study. Subjects were randomly assigned into two groups which are treatment and control group. For a 3 months period, the treatment group was given 2x100 g soursop fruit juice per day and the control group was left without treatment.

Blood pressure was measured by medical team using Omron HEM-907 (digital automatic blood pressure monitoring) every 2 weeks (3 times readings for each) in each subject's home. Subjects were examined in sitting position. Evaluation of laboratory examination was taken at week 0, 7 and 13.

ELIGIBILITY:
Inclusion Criteria:

1. pre-hypertensive patients in accordance with JNC 7 (Joint National Committee 7) criteria,
2. male or female resident in Mlati, Sleman with or without family history of hypertension,
3. age 30-59 years,
4. high normal uric acid levels (≥ 5 and < 7 mg/dL) and
5. agreed to follow the study by giving their informed consent.

Exclusion Criteria:

1. have a history of diabetes, chronic renal failure,
2. using hormonal contraceptive,
3. in pregnancy,
4. taking uric acid-lowering drugs (allopurinol, probenecid),
5. positive urine reduction, positive proteinuria, creatinine > 1.5 g/dL, Blood Glucose > 126 g/dL.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Change in baseline morning home blood pressure at week 7 and 13 | Week 0, 7 and 13
  Blood pressure was measured by medical team using Omron HEM-907 (digital automatic blood pressure monitoring) every 2 weeks (3 times readings for each) in each subject's home. Subjects were examined in sitting position.
Change in baseline serum uric acid at week 7 and 13 | Week 0, 7 and 13
  Blood sample was taken to measure serum uric acid level

SECONDARY OUTCOMES:
Change in baseline CKD-Epi at week 7 and 13 | Week 0, 7 and 13
  Measurement of glomerular filtration rate
Change in baseline uric acid excretion at week 7 and 13 | Week 0, 7 and 13
  24-h urine sample was taken to measure uric acid excretion

CONTACTS AND LOCATIONS:
Overall Officials: Mochammad Sja'bani, PhD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, University of Gadjah Mada
Locations (1):
- Mlati 2 Health Center working area (Sumberadi, Tlogoadi,Tirtoadi), Sleman, Special Region of Yogyakarta, Indonesia